CLINICAL TRIAL: NCT07180433
Title: Piloting 18F-FAPI PET/MRI for Applications in Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 639856/23
Record Dates: First submitted 2025-06-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FAPI-PET/MRI (Experimental): The patients will be injected 2 MBq/kg 18F-FAPI, prior to PET/MRI acquisition
  Interventions: Diagnostic Test: FAPI PET/MR

INTERVENTIONS:
Diagnostic Test: FAPI PET/MR — The patients will be injected intravenously with 2 MBq/kg 18F-FAPI, 60 minutes before the PET/MRI acquisition. The PET/MRI examinations will be performed on a Siemens Biograph mMR (Siemens Healthcare, Erlangen, Germany) with software version VE11P. Static PET will be acquired simultaneously with MRI using two protocols; a one bed position protocol in prone position covering the breast and a whole body 4-5 bed position protocol in supine position covering brain to thighs. Total acquisition time of the breast protocol will be approximately 20 minutes. Total acquisition time of the whole-body protocol will be approximately 30 minutes.

SUMMARY:
Breast cancer is the most common type of cancer in Norwegian women, with 4,224 new cases in 2022. More precise diagnosis are expected to result in more accurate assessment of treatment effect, and to contribute to both providing better treatment and reducing overtreatment. Fibroblast activating protein (FAP) is expressed in the tumor stroma of 90% of all epithelial-based tumors, including breast tumors. Inhibitors for this protein (FAPI) has been developed for use as radioactive tracers. Breast tumors of various histopathological types, and local metastatic lymph nodes, have shown high uptake for such tracers. The main aim of this project is to establish 18F-FAPI PET/MRI for use in breast cancer in a wide range of disease stages. We will evaluate how FAPI PET/MRI correlates with histopathological assessment, the method's ability to grade tumors - including assessment of treatment - compared to CT, scintigraphy and FDG PET/CT, and ability to detect local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are accepting to undergo 18F-FAPI PET/MRI examinations and

  1. diagnosed with local invasive breast cancer,
  2. scheduled for neoadjuvant therapy as primary treatment,
  3. has recurrent or new breast cancer, or
  4. scheduled for neoadjuvant therapy as primary treatment with FDG-PET/CT applied for staging.

Exclusion Criteria:

* other primary malignancies than breast cancer, renal insufficiency or know allergy towards contrast agents, and MR incompatible implants.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 18F-FAPI-PET/MRI in detection of breast cancer lesions | Baseline
  Diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of 18F-FAPI-PET/MRI in detecting breast cancer lesions, including primary tumors, regional lymph node metastases, distant metastases, and local/distant recurrences. Interpretation will be based on consensus assessment by nuclear medicine physicians and radiologists. Histopathology and/or conventional imaging (CT, FDG-PET, bone scintigraphy) will serve as the reference standards.

SECONDARY OUTCOMES:
Correlation of standardized uptake values of 18F-FAPI to histologically proven characteristics of the breast cancer lesions | Baseline
  Quantitative PET compared to standard histopathology of breast tumours and axillary lymph nodes, including number and size, grading, receptor status, and histological type
Diagnostic accuracy of 18F-FAPI PET/MR compared to MR only in prediction/evaluation of response to neoadjuvant chemotherapy | From baseline to surgery (~3-6 months)
  PET/MRI data compared to clinical response to chemotherapy (cR), pathologic complete response (pCR) and residual cancer burden (RCB)
Diagnostic accuracy of 18F-FAPI PET/MR compared to standard CT/bone scintigraphy in staging of breast cancer | Baseline
  Comparison of detection rates by PET/MR data to standard CT/bone scintigraphy.
Diagnostic accuracy of 18F-FAPI PET/MR compared to CT/bone scintigraphy in detection of recurrence. | Baseline
  Comparison of detection rates by PET/MR data to standard CT/bone scintigraphy.
Diagnostic accuracy of 18F-FAPI PET/MR compared to 18F-FDG PET/CT. | Baseline
  Comparisons of consesus readings by radiologists and nuclear medcine physisians.